

## Hemodynamic Effect of Norepinephrine Versus Vasopressin on the Pulmonary Circulation in Cardiac Surgery Patients: a Comparative- effectiveness Pragmatic Trial

10/04/2024

NCT Identifier: NCT04501861, registered on August 6<sup>th</sup>, 2020



## PATIENT INFORMATION SHEET

## Hemodynamic Effect of Norepinephrine Versus Vasopressin on the Pulmonary Circulation in Cardiac Surgery Patients: a Comparative- effectiveness Pragmatic Trial

## Dear Patient:

This letter describes a research project in which you may be enrolled. This project is approved by the Cleveland Clinic Institutional Review Board.

During your upcoming cardiac surgery, your anesthesiologist may use several medications to support your blood pressure, to make surgery as safe as possible for you. Two medications we commonly use to support the blood pressure are 1) norepinephrine and 2) vasopressin. In our current practice at the Cleveland Clinic, each individual anesthesiologist chooses which, or both, of these to use. Our group uses these drugs interchangeably, which does not deviate from the standard of cardiac anesthesia and surgical care.

We know that both norepinephrine and vasopressin work similarly to support the blood pressure during surgery. We are conducting this investigation to see if either of those commonly used drugs has any more effect than the other on the blood vessels in your lungs. In order to do so, we will be using one of those drugs preferentially over the other. If the one drug is not enough to support your blood pressure safely, additional medications will be used as our primary goal is to make this as safe as we can for you during your surgery. Since the trial is not "blinded", both your anesthesiologist and your surgeon will know which medication (norepinephrine or vasopressin) you will receive. **This investigation will not change any other aspect of your care**, and you will otherwise receive exactly the standard of care for your anesthesia and surgery. If there is any reason your anesthesiologist to believe that one medication is better for your particular case than the other, you will not be enrolled in the study, and you will receive the medication which is believed to be safest for you. In case you do not require these two medications during surgery, you will not be included in the study.

Information such as your name, day of surgery, type of surgery, surgical data, vital signs during surgery, laboratory tests and related complications, will be collected from your medical record during your surgery. All data will be securely stored and kept confidential and only the investigators will have access to it. Knowledge gained from this investigation will ultimately improve patient care and benefit future patients.



If you have any questions about the investigation or would **prefer NOT to be included**, please inform us by calling one of our cell phone numbers or sending an email, and you will be able to contact one of the investigators directly. When you choose to opt out from the investigation, your anesthesia team will be informed that you are not part of the investigation, and no data will be collected during your surgery and hospital stay.